CLINICAL TRIAL: NCT02948374
Title: Biomarkers in Cerebrospinal Fluid in Critical Care Patients With Delirium
Acronym: BIO-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Lundin, Professor, Sahlgrenska University Hospital
Other Study IDs: LUA-74202
Record Dates: First submitted 2016-09-09; First posted 2016-10-28 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Delirium; Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delirium positive: Patients with a positive CAM-ICU test
- Delirium negative: Patient without delirium determined with the CAM-ICU test

SUMMARY:
Critical care patients are at a high risk of developing delirium and impaired cognitive function 3 and 12 months after their ICU stay. In this study the aim is to try to elucidate the pathophysiology behind delirium in the ICU and subsequent development of cognitive dysfunction in ICU survivors.

Biomarkers in cerebrospinal fluid (CSF) will be analysed in patients with and without delirium in the ICU. Samples will also be taken 3 and 12 months after the ICU-stay. CSF will also be obtained in healthy age- and sexmatched controls undergoing surgery.

DETAILED DESCRIPTION:
Critical care patients are at a high risk of developing delirium, a form of acute brain dysfunction, and may develop impaired cognitive function 3 and 12 months following their ICU stay.

In this study the aim is to try to elucidate the pathophysiology behind delirium in the ICU comparing patients with and without delirium and possible development of cognitive dysfunction in ICU survivors. Neuroinflammatory markers and markers of structural damage in cerebrospinal fluid (CSF) will be analysed in patients with and without delirium assessed with the CAM-ICU (Confusion Assessment Method) test in the ICU. CSF samples will also be taken in ICU-survivors, 3 and 12 months after the ICU-stay. For comparison CSF will be obtained in healthy age- and sexmatched controls undergoing surgery in spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU for acute respiratory, septic and/or circulatory chock

Exclusion Criteria:

* Abnormal coagulation
* Recent exposure to intensive care
* Patients unable to assess for delirium
* Patients difficult to follow up
* Patients expected to live less than 24 hrs
* Patients with known cognitive dysfunction based on medical records or relatives report
* Abnormal coagulation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of biomarkers for inflammation and structural damage in the cerebrospinal fluid in patient with or without delirium in the ICU | At Baseline samples of CSF are taken in patients evaluated with CAM-ICU test and with EEG for the presence or absence of delirium
  Delirium in the ICU is assessed with the CAM-ICU test and by EEG in patients admitted to the ICU for respiratory failure or circulatory or septic chock

SECONDARY OUTCOMES:
Concentration of neuroinflammatory biomarkers and markers of neural damage in the cerebrospinal fluid in surviving patients with and without cognitive dysfunction 3 months after their ICU stay. | Three months after the patients have left the intensive care unit samples of CSF will be taken in surviving patients in the Outcome 1 group above.
Concentration of neuroinflammatory biomarkers and markers of neural damage in the cerebrospinal fluid in surviving patients with and without cognitive dysfunction 12 months after their ICU stay. | Twelve months after the patients have left the intensive care unit samples of CSF will be taken in surviving patients in the Outcome 1 group above.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lundin, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No